CLINICAL TRIAL: NCT01157325
Title: Comparison of the Cesarean Rate Between Parturients Who Received Neuraxial Analgesia and Those Who Did Not
Brief Title: Cesarean Rate in Parturients Without Neuraxial Analgesia
Acronym: CRINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NJMU10-201; NJFY2010Y116 (Other Grant/Funding Number: Nanjing Maternity and Child Health Care Hospital)
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Labor
Keywords: Epidural analgesia; Latent analgesia; Active analgesia; Cesarean section

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-neuraxial analgesia (Active Comparator): Parturients will not receive neuraxial analgesia
  Interventions: Procedure: Non-neuraxial analgesia
- Neuraxial analgesia (Active Comparator): Parturients will receive neuraxial analgesia
  Interventions: Procedure: Neuraxial analgesia

INTERVENTIONS:
Procedure: Neuraxial analgesia — Neuraxial analgesia will be given at any time if the parturient requested analgesia
  Arms: Neuraxial analgesia
Procedure: Non-neuraxial analgesia — No neuraxial analgesia will be given to those who will not want to an analgesia
  Arms: Non-neuraxial analgesia

SUMMARY:
Currently, it is certain that neuraxial analgesia in early stage of labor and delivery dose not increase the risk of Cesarean section. However, given ethical reasons, whether such a medical procedure could increase the Cesarean rate compared with those who did not received neuraxial analgesia or not is yet to be known. It is difficult to perform such a study in occidental countries because they have a higher rate of labor analgesia. On the contrary, the rate of labor analgesia in China is up to date only 1%, so it can be done easily. The investigators hypothesized that no neuraxial analgesia itself were a risk factor to Cesarean section. Therefore, the investigators design this study to compared the effect of neuraxial analgesia on the rate of Cesarean delivery with those who did not received neuraxial analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 19yr, <=40 yr
* Height 140 - 170 cm
* Singleton pregnancy
* Uncomplicated pregnancy
* Chinese

Exclusion Criteria:

* Multiple gestations
* Pregnancy-induced hypertension
* Diabetes mellitus
* Chronic pain
* Allergic to opioids and/or local anesthetics
* Failed to performing inter lumbar space catheterization
* Organic dysfunction
* Contraindications for neuraxial analgesia

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Cesarean rate | One day after birth
  Rate of Cesarean delivery in both neuraxial and non-neuraxial analgesia women

SECONDARY OUTCOMES:
Instrumental delivery | One day after birth
  The rate of instrument-assisted delivery in both neuraxial and non-neuraxial analgesia women
VAS pain intensity | At the begining of labor (0 min)
  Labor pain intensity assessed using visual analog scale (VAS)
VAS pain intensity | At the cervix 10 cm (This time may be subjected to change in different patients)
  Labor pain intensity assessed using visual analog scale (VAS)
VAS pain intensity | 2h after cervix 10 cm
  Labor pain intensity assessed using visual analog scale (VAS)
Time of successful labor | From the initial of labor (0 min) to completion of delivery (this is changable individually)
  Labor duration in both neuraxial and non-neuraxial analgesia women
Time of the first stage of labor | From initial of the labor to the cervix reached to 10 cm (Different in different patients)
  Duration of the first stage of labor
Time of second stage of labor | From the cervix at 10 cm to successful delivery of the baby (this is changable individually)
  Duration of the second stage of labor
Overall feeling of satisfaction of the labor | At the end of successful baby delivery (it is changable individually)
  Satisfaction assessed using a visual analog scale (VAS) at the end of the labor delivery
Side effects | From the initial of labor (0 min) to the end of the labor (is is changable individually)
  Side effects recorded from the labor initiation to successful delivery

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, MPH, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China